CLINICAL TRIAL: NCT03590405
Title: Uterus Transplantation LD - Feasibility Study - Sahlgrenska - Bellevue Medical Centre
Brief Title: Uterus Transplantation LD - Feasibility Study - Sahlgrenska - BMC
Acronym: GOT-BMC-UTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Saint Joseph University, at Bellevue Medical Centre (Unknown)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sahlgrenska-BMC-UTx
Record Dates: First submitted 2018-06-17; First posted 2018-07-18 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Mrk Anomaly; Infertility, Female
Keywords: uterus; infertility; transplantation
MeSH Terms: conditions — Mullerian aplasia; Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uterus transplantation (Experimental): uterus transplantation from living donor with the donor being close relative
  Interventions: Procedure: uterus transplantation surgery and IVF

INTERVENTIONS:
Procedure: uterus transplantation surgery and IVF — IVF before surgery living donor uterus transplantation ET

SUMMARY:
Medical know-how concerning uterus transplantation will be transferred to new site by structured process involving theory, animal workshops and a clinical feasibility study on human subjects.

DETAILED DESCRIPTION:
Medical know-how concerning uterus transplantation will be transferred to new site by structured process involving theory, animal workshops and surgery.

Theory and common animal workshops have been ongoing for 3 years. The team from Bellevue Medical Centre is affiliated to St Joseph, University, Beirut

ELIGIBILITY:
Inclusion criteria recipient

* age < 38 years
* psychologicaly stable
* BMI < 35
* no systemic disease
* no standing medication
* in a stable relationship or married
* normal ovarian reserve
* absolute uterine factor infertility
* normal kidney function

Inclusion criteria donor

* close relative to recipient
* age < 60 years
* normal pregnancies
* maximum two cesarean sections
* BMI < 35
* no major systemic disease
* no previous major surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females
Enrollment: 2 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
live birth | 3 years
  live birth

CONTACTS AND LOCATIONS:
Overall Officials: Mats Brännström, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Mats Brännström, Gothenburg

IPD SHARING:
Plan to Share IPD: No